CLINICAL TRIAL: NCT01965366
Title: A Pilot Study of the Effects of Dexamethasone Administration on Virtual Reality Exposure Therapy for PTSD
Brief Title: Dexamethasone Plus Virtual Reality Exposure Therapy for PTSD
Acronym: Dex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor in Psychiatry, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00068205
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: PTSD
Keywords: Dexamethasone; Virtual Reality; Military; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Virtual Reality Exposure Therapy; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone + VRE (Active Comparator): 0.5 mg DEX + virtual reality exposure therapy
  Interventions: Behavioral: Virtual reality exposure therapy; Drug: 0.5 mg DEX
- Placebo + VRE (Placebo Comparator): Placebo + virtual reality exposure therapy
  Interventions: Behavioral: Virtual reality exposure therapy

INTERVENTIONS:
Behavioral: Virtual reality exposure therapy — Virtual reality exposure (VRE) therapy is a form of exposure therapy in which participants are helped to confront their traumatic memories in a therapeutic manner. They describe the events out loud and their therapist attempts to match what they are describing in the virtual reality. This is done repeatedly, allowing distress associated with these memories to decrease. Material that emerges during the VRE exposure is processed, or discussed, after the exposure, allowing participants to think about themselves and the event differently.
Drug: 0.5 mg DEX — A dose of DEX will be given the night before (approximately 10 hours before) each of 5 to 11 individual virtual reality exposure (VRE) therapy sessions.
  Other Names: Dexamethasone
  Arms: Dexamethasone + VRE

SUMMARY:
Evidence from preliminary studies suggests that people with PTSD have heightened fear responses and that cortisol suppression reduces this heightened fear. Research has shown the drug dexamethasone (DEX), a cortisol suppressor, reduces the startle response in civilians with PTSD. This current research proposal represents a blinded, randomized, placebo-controlled efficacy study with the goal of determining whether a drug that suppresses the stress hormone cortisol will increase the efficacy of exposure therapy. Specifically, it is proposed that a dose of DEX, given the night before (approximately 10 hours before) each of 5 to 11 individual virtual reality exposure (VRE) therapy sessions, will significantly enhance the rate of response and possibly the efficacy of treatment. Participants will be treated until they have experienced at least a 70% reduction in PTSD symptoms from baseline or up to 12 sessions or until they and their therapist agree treatment should be terminated, a minimum of 6 sessions to a maximum of 12 sessions. Comprehensive multi-modal outcomes will be assessed by independent assessors blind to subject condition on interviews, self-report measures, and psychophysiological measures. Participants will be assessed pre- and post-treatment and at a follow-up of 3, 6 and 12 months to assess long term effects.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 60 males and females between ages of 21 and 65.
2. Participants must meet DSM-V criteria for PTSD due to exposure to a trauma while serving in Operation Iraqi Freedom and/or Operation Enduring Freedom-Afghanistan and Operation New Dawn.
3. Patients must be literate in English.
4. Patients must be medically healthy or medically stable such that the stress of VR and DEX are not contraindicated.
5. Participants must comprehend his or her role in the study and the risks involved in order to be entered.

Exclusion Criteria:

1. Patients with a history of mania, schizophrenia, or other psychoses;
2. Patients with prominent suicidal ideation;
3. Patients with current alcohol or drug dependence;
4. Patients unable to tolerate wearing the VR helmet;
5. Patients unwilling to take study medication;
6. Patients on psychotropic medication(s) must have been on a stable dose for at least 2 weeks prior to beginning the study and must agree not to change their current medication regimen throughout the course of the study. The concomitant use of psychotropic medications will be recorded and examined in data analyses.
7. Patients with special medical conditions such as pregnancy, renal insufficiency, or a history of significant head injury
8. Active medical disorders contributing to psychiatric sx e.g. hypo or hyperthyroidism, SLE, advanced cirrhosis, etc. (per clinical judgment of study physician)
9. Patients stabilized on potentially data-obscuring medications (glucocorticoids).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10; Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rothbaum, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone + VRE | Placebo + VRE
Started | 13 | 14
Completed | 3 | 9
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone + VRE | Placebo + VRE | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 5 | 5 | 10
  black | 5 | 7 | 12
  other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in The Clinician Administered PTSD Scale (CAPS)Scores
Description: The Clinician Administered PTSD Scale (CAPS) provides a diagnostic measure of PTSD and a continuous measure of the severity, frequency, and intensity of the three symptom clusters (intrusion, avoidance, and arousal) and overall PTSD. The assessor combines information about frequency and intensity of an item into a single severity rating. Severity Rating: 0. Absent; 1. Mild / subthreshold;2. Moderate / threshold; 3. Severe / markedly elevated; 4.Extreme / incapacitating. The assessor combines information about frequency and intensity of an item into a single severity rating. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Scores may range from 0-80, with a higher score indicating more reported symptoms of PTSD.
Time Frame: Baseline and immediate post treatment (up to 12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone + VRE | Placebo + VRE
Number analyzed (Participants) | 3 | 9
units on a scale | -11 (10.44) | -15.22 (12.40)

2. Secondary Outcome: Change in The PTSD Symptom Scale Scores
Description: The PTSD Symptom Scale (PSS) is a 17-item interview used to aid in the detection and diagnosis of PTSD. The structure and content of the PSS mirror the DSM-IV criteria for PTSD. For each item, the interviewer assigns a rating to reflect a combination of frequency and severity (from O = "not at all" to 3 = "5 or more times per week/very much"). Scores range from 0-51, with higher scores indicating more reported symptoms of PTSD. A score of 13 or higher indicates the likelihood of PTSD.
Time Frame: Baseline and immediate post treatment (up to 12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone + VRE | Placebo + VRE
Number analyzed (Participants) | 3 | 9
units on a scale | -9 (16.97) | -16.65 (12.69)

ADVERSE EVENTS:
Time Frame: 12 months of follow up
Arm/Group | Dexamethasone + VRE | Placebo + VRE
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT01965366/Prot_SAP_000.pdf